CLINICAL TRIAL: NCT05829031
Title: Tailored Ecological Momentary Music Intervention to Reduce Stress in the Daily Life of Turkish Immigrant Women
Brief Title: Tailored Ecological Momentary Music Intervention for Stress Reduction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The anticipated study duration was two years. Despite sustained recruitment efforts, the required number of eligible participants could not be enrolled within this timeframe. Therefore, the study was terminated.
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Urs Nater, Professor, University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMMI-T Main
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-03

CONDITIONS: Stress, Psychological; Stress, Physiological; Discrimination, Racial
Keywords: Ecological Momentary Intervention; Music; Stress reduction; Discrimination; Cortisol; Alpha-Amylase
MeSH Terms: conditions — Stress, Psychological; Racism

STUDY DESIGN:
Intervention Model Description: Intra-individually randomized design: Participants will be randomly assigned (50:50) to either the intervention condition or the control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Music listening vs. No music listening (Experimental): Every participant will be randomly assigned (50:50) to one of the following two conditions: Music listening after a stressful and/or discriminatory event (i.e., intervention condition) or no music listening after a stressful and/or discriminatory event (i.e., control condition).
  Interventions: Behavioral: Targeted music listening

INTERVENTIONS:
Behavioral: Targeted music listening — Participants listen to self-selected relaxing music. They can choose between a duration of either 10 minutes or 20 minutes.

SUMMARY:
Ethnic discrimination is associated with mental and physical health impairments. In view of the negative impact of discrimination on health, it is of great importance to investigate interventions to counteract these negative effects.

Based on findings of a pilot study (clinicaltrials.gov identifier: NCT04957966), this study investigates the effectiveness of a tailored ecological momentary music intervention to reduce biological (salivary cortisol, salivary alpha-amylase) and psychological (perceived stress, perceived ethnic discrimination) stress reactions after discriminatory and/or stressful events in the daily life of Turkish immigrant women (N = 50, age range 18-65 years).

An intra-individually randomized design will be used, i.e., participants will be assigned on a random basis either to intervention events (they can choose to listen to music for the duration of 10 or 20 minutes) or to control events (participants are instructed to not listen to music). The whole study period consists of 35 days with a baseline period (week 1), intervention period (week 2-4), and post period (week 5).

DETAILED DESCRIPTION:
Ethnic discrimination (ED) represents a complex stressor that triggers psychobiological stress reactions (Pascoe & Smart Richman, 2009). Experienced chronically, ED can adversely affect mental and physical health (e.g., Lewis et al., 2015; Schmitt et al., 2014), most likely due to dysregulations of psychobiological stress systems (Chrousos, 2009; Schlotz, 2019). In this regard, women may be particularly affected as they face discrimination based on both ethnicity and gender more often compared to men (e.g., Harnois, 2014; Seaton & Tyson, 2019). Considering the resulting health impairments, it is of great importance to investigate strategies that can mitigate the occurring stress reactions and thereby contribute to health promotion. Therefore, we conducted a pilot study to test the feasibility of an ecological momentary music intervention aiming to reduce stress levels of affected individuals (clinicaltrials.gov identifier: NCT04957966). Based on the findings of the pilot study and power calculations, we will now conduct a larger main study. The primary aim of our study is to examine the effectiveness of an ecological momentary music intervention to reduce psychological and biological (cortisol, alpha-amylase) stress levels after stressful and/or discriminatory events in the daily life of chronically discriminated Turkish immigrant women.

We hypothesize that listening to self-selected, relaxing music after an event of acute stress and/or ethnic discrimination in daily life will result in stronger decreases of psychological (perceived stress, perceived ethnic discrimination) and biological (cortisol, alpha-amylase) stress levels compared to no music listening (immediate effect). Further, we expect a decrease in diurnal psychological and biological stress levels throughout the study period (intermediate effect).

The study consists of three phases: Baseline phase (week 1), intervention phase (week 2 to 4), post intervention phase (week 5).

During the baseline and post intervention phase, we will assess participants' psychological and biological stress fluctuations and perceived ethnic discrimination in daily life. Therefore, participants will be prompted three times a day (11:00 am, 3:00 pm, 7:00 pm) through a study app to answer questions on their momentary levels of stress, perceived discrimination, positive and negative affect, and their music-listening activities (time-contingent data entries). Additionally, whenever a stressful and/or discriminatory event occurs, participants will be instructed to initiate a data entry by themselves in order to report their momentary levels of stress, perceived discrimination, positive and negative affect, and to answer questions on the current situation. To investigate activities after such self-initiated, event-contingent data entries, the app will prompt the participants 20 minutes later for an additional data entry (post). As part of every time-contingent and event-contingent report, participants will provide a saliva sample for the analysis of biological stress markers: salivary cortisol levels as index of hypothalamic-pituitary-adrenal axis (HPA axis) activity, salivary alpha-amylase as index of autonomic nervous system (ANS) activity.

Every evening before going to bed, participants will complete a daily diary assessment via the study app. In this diary, participants will be asked about their current perceived stress, perceived discrimination, positive and negative affect, fatigue, and coping strategies. Additionally, they will be asked whether discriminatory or stressful events had happened over the course of the day and if so, to describe the event(s). This data entry will not require the collection of a saliva sample.

During the intervention phase (week 2 to 4), the sampling protocol will be the same as in the baseline and post intervention phase (i.e., time-contingent data entries, daily diary assessment, self-initiated event-contingent data entries, post). Additionally, participants will be randomly assigned (50:50) to either the intervention condition (listening to self-selected, relaxing music; participants can choose between the duration of 10 or 20 minutes) or the control condition (no music listening; participants are instructed to continue their pre-data entry activities) after every self-initiated event-contingent report. This intra-individually randomized study design will allow us to compare the effects of music listening vs. no music listening after stressful/discriminatory events on psychological and biological stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Turkish immigrants (1st or 2nd generation)
* Chronic ethnic discrimination (value of or above 104 on the Everyday Discrimination Scale)
* 18-65 years
* sex: female

Exclusion Criteria:

* Insufficient proficiency of the German language
* Body mass index (BMI) above 30 kg/m2
* Schizophrenia
* Substance-induced disorder in the past 2 years
* Chronic somatic diseases
* Medical conditions or medications known to affect endocrine or autonomic functioning
* Abuse of alcohol in the past 6 months
* Drug use in the past year, cannabis use in the past 14 days
* Pregnancy
* Breastfeeding
* Impaired hearing or absolute pitch

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Stress Experience | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: 20 minutes after T0
  Momentary stress level: visual analogue scales (VAS; 0-100, higher scores indicate a greater level of momentary stress)
Change in Short-Term Neuroendocrine Stress: Hypothalamic-Pituitary-Adrenal Axis | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: 20 minutes after T0
  Biological Marker: Salivary Cortisol
Change in Short-Term Neuroendocrine Stress: Autonomic Nervous System | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: 20 minutes after T0
  Salivary Alpha-Amylase

SECONDARY OUTCOMES:
Change in positive and negative affect | from baseline period (week 1) to post period (week 5)
  PANAS (Positive Affect Negative Affect Scale; Watson et al., 1988; German version by Krohne et al., 1996) is a self-report questionnaire that consists of two scales to measure positive affect and negative affect, each scale consists of 10 items (5-point Likert Scales, for every scale higher scores indicate greater positive/negative affect)
Change in fatigue | from baseline period (week 1) to post period (week 5)
  5 items (one of each scale) of the MFI (Multidimensional Fatigue Inventory; Smets et al., 1995), a self-report questionnaire consisting of 20 items that are assigned to 5 scales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation (5-point Likert Scales, higher scores on each subscale indicate greater levels of each subscale-specific type of fatigue)
Change in coping behavior | from baseline period (week 1) to post period (week 5)
  5 items of the Brief-COPE (Coping Orientation to Problems Experienced Inventory; Carver, 1997; German version by Knoll et al., 2005), a self-report questionnaire that consists of 28 items to measure effective and ineffective ways of coping with stressful life events; one item of each subscale: active coping, use of emotional support, use of instrumental support, venting, religion; 5-point Likert-Scales with higher scores for each subscale indicating a greater level of the subscale-specific coping behavior)
Change in avoidance behavior regarding discriminatory events | from baseline period (week 1) to post period (week 5)
  Combination of the following 4 items to measure change in avoidance behavior:
  * 3 items of the avoidance subscale of the CSI (Coping Strategy Indicator; Amirkhan, 1990), a self-report questionnaire of situational coping that consists of 33 items with the subscales avoidance, problem solving, and seeking social support (5-point Likert-Scales with higher scores indicating greater levels of avoidance behavior)
  * one self-developed item to measure avoidance behavior, in particular the item measures if the person avoided situations and/or persons for fear of being discriminated against (5-point Likert-Scales with higher scores indicating greater levels of avoidance behavior)
Change in anticipation of discriminatory events | from baseline period (week 1) to post period (week 5)
  3 items of the Racism-related Vigilance Scale (Clark et al., 2006), a 6-item scale to measure heightened vigilance regarding discriminatory events (5-point Likert-Scales with higher scores indicating greater levels of anticipation of discriminatory events)
Perceived burden regarding the intervention | after 5 weeks
  10 items of a self-developed questionnaire on perceived burden regarding the intervention (5-point Likert Scales, higher scores indicate greater levels of perceived burden)
Satisfaction with the intervention | after 5 weeks
  6 items of a self-developed questionnaire on satisfaction with the intervention (5-point Likert Scales, higher scores indicate greater levels of satisfaction)
Usage Rate of the App | after 5 weeks
  Timestamped log-data of the app to determine usage rate by the participants (higher usage rate indicates a greater feasibility of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Ricarda Nater-Mewes, Dr. Dr., Principal Investigator — University of Vienna; Urs Nater, Prof., Principal Investigator — University of Vienna
Locations (1):
- University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request.

REFERENCES:
- [Background] Amirkhan JH. A Factor Analytically Derived Measure of Coping - the Coping Strategy Indicator. J Pers Soc Psychol 1990;59:1066-74.
- [Background] Chrousos GP. Stress and disorders of the stress system. Nat Rev Endocrinol. 2009 Jul;5(7):374-81. doi: 10.1038/nrendo.2009.106. Epub 2009 Jun 2. PMID 19488073
- [Background] Clark R, Benkert RA, Flack JM. Large arterial elasticity varies as a function of gender and racism-related vigilance in black youth. J Adolesc Health. 2006 Oct;39(4):562-9. doi: 10.1016/j.jadohealth.2006.02.012. Epub 2006 Jul 10. PMID 16982392
- [Background] Harnois CE. Are perceptions of discrimination unidimensional, oppositional, or intersectional? Examining the relationship among perceived racial-ethnic-, gender-, and age-based discrimination. Sociol Perspect 2014;57:470-87.
- [Background] Knoll N, Rieckmann N, Schwarzer R. Coping as a mediator between personality and stress outcomes: A longitudinal study with cataract surgery patients. Eur J Pers 2005;19:229-47.
- [Background] Krohne HW, Egloff B, Kohlmann C-W, Tausch A. Untersuchungen mit einer deutschen Version der
- [Background] Lewis TT, Cogburn CD, Williams DR. Self-reported experiences of discrimination and health: scientific advances, ongoing controversies, and emerging issues. Annu Rev Clin Psychol. 2015;11:407-40. doi: 10.1146/annurev-clinpsy-032814-112728. Epub 2015 Jan 2. PMID 25581238
- [Background] Pascoe EA, Smart Richman L. Perceived discrimination and health: a meta-analytic review. Psychol Bull. 2009 Jul;135(4):531-54. doi: 10.1037/a0016059. PMID 19586161
- [Background] Schlotz W. Investigating associations between momentary stress and cortisol in daily life: What have we learned so far? Psychoneuroendocrinology. 2019 Jul;105:105-116. doi: 10.1016/j.psyneuen.2018.11.038. Epub 2018 Nov 27. PMID 30503527
- [Background] Schmitt MT, Branscombe NR, Postmes T, Garcia A. The consequences of perceived discrimination for psychological well-being: a meta-analytic review. Psychol Bull. 2014 Jul;140(4):921-48. doi: 10.1037/a0035754. Epub 2014 Feb 17. PMID 24547896
- [Background] Seaton EK, Tyson K. The Intersection of Race and Gender Among Black American Adolescents. Child Dev. 2019 Jan;90(1):62-70. doi: 10.1111/cdev.13093. Epub 2018 May 19. PMID 29777539
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Derived] Hirsch S, Nater UM, Mewes R. Smartphone-based ecological momentary music intervention to reduce stress in Turkish immigrant women: protocol. BMJ Open. 2025 Apr 5;15(4):e090518. doi: 10.1136/bmjopen-2024-090518. PMID 40187786
- See also: clinicaltrials.gov registration of the corresponding pilot study — https://clinicaltrials.gov/ct2/show/NCT04957966?term=EMMI-T&draw=2&rank=1